CLINICAL TRIAL: NCT01410838
Title: Effects of Ingesting Monosodium Glutamate (MSG) on Energy Balance and Eating Behavior Following Moderate Energy Restriction and Weight Loss in Overweight Women
Brief Title: Effects of Monosodium Glutamate on Energy Balance and Eating Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Ajinomoto USA, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WHNRC 222718-2
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Weight Gain; Food Preferences
Keywords: Obesity; Food preferences; Eating Behavior
MeSH Terms: conditions — Obesity; Weight Gain; Food Preferences; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Broth- NaCl (Placebo Comparator): Sodium chloride containing broth matched for sodium content to the MSG broth
  Interventions: Other: Broth
- Broth- MSG (Active Comparator): MSG containing broth with the same sodium content as the placebo comparator.
  Interventions: Other: Broth

INTERVENTIONS:
Other: Broth — 200 mL of sodium chloride containing broth, consumed three times per day
  Arms: Broth- NaCl
Other: Broth — 200 mL of MSG containing broth consumed three times per day
  Arms: Broth- MSG

SUMMARY:
This study will test whether regular consumption of Monosodium Glutamate (MSG) immediately prior to each of the three major meals (breakfast, lunch, dinner) inhibits body weight and fat regain following a period of moderate, yet clinically significant weight loss.

DETAILED DESCRIPTION:
The proposed study enables us to assess the long term effects of consuming MSG on body weight regain following weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 19-45
* BMI 27-35
* Blood pressure <140/90
* Non-smoking

Exclusion Criteria:

* Anemic: hgb < 11.5 mg/dL
* Sensitivity to MSG (self reported)
* Pregnant or planning to get pregnant
* Taking medication for hypertension, depression, or weight loss
* Diabetic
* Vegetarian
* MRI Contraindications: internal metal, braces on teeth, history of metal in the eye, claustrophobia
* blindness or heavily corrected vision
* not fluent in English

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in body weight | weeks 11, 12, and 25
  Subjects will have their body weight measured to determine the effect of MSG on body weight regain following weight loss.

SECONDARY OUTCOMES:
Change in body fat | weeks 11 and 25
  Volunteers will have their body fat measured by DEXA (Dual X-ray Absorptiometry) to determine the effect of MSG on body fat regain following weight loss.
Change in eating behavior | weeks 11, 12 and 25
  The effect of MSG on eating behavior will be measured using questionnaires, sensory evaluation testing, stress responsivity, and liking and wanting tests, and appetite assessments.
Change in resting energy expenditure | weeks 11, 12, and 25
  The effect of MSG on resting energy expenditure will be measured using respiratory gas exchange using a metabolic cart system.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Laugero, PhD, Principal Investigator — WHNRC, ARS, University of California Davis
Locations (1):
- Western Human Nutrition Center, University of California Davis, Davis, California, United States

REFERENCES:
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/Main/docs.htm?docid=11240